CLINICAL TRIAL: NCT01543074
Title: Dietary Histone Deacetylase (HDAC) Inhibitors
Brief Title: Dietary Histone Deacetylase Inhibitors (HDAC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Roderick Dashwood, Director Center for Epigenetics & Disease Prevention, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CA122959
Record Dates: First submitted 2012-02-17; First posted 2012-03-02 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Histone Deacetylase (HDAC) Activity
Keywords: HDAC; histone acetylation; broccoli sprout extract; garlic oil; PBMCs
MeSH Terms: conditions — Motor Activity | interventions — allyl sulfide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BSE placebo & garlic oil placebo (Placebo Comparator): Two BSE placebo capsules and one garlic oil placebo capsule per day for seven days
  Interventions: Dietary Supplement: BSE placebo; Dietary Supplement: Garlic Oil Placebo
- garlic oil plus BSE placebo (Active Comparator): one garlic oil capsule plus 2 BSE placebo capsules per day for seven days
  Interventions: Dietary Supplement: BSE placebo; Dietary Supplement: Garlic oil
- BSE plus garlic oil placebo (Active Comparator): two BSE capsules plus one garlic oil placebo capsule per day for seven days
  Interventions: Drug: BSE; Dietary Supplement: Garlic Oil Placebo
- BSE & Garlic Oil (Active Comparator): two BSE and one garlic oil capsule per day for seven days
  Interventions: Dietary Supplement: Garlic oil; Drug: BSE

INTERVENTIONS:
Dietary Supplement: BSE placebo — 2 pills = 0 micromoles of Sulforaphane/day
  Other Names: Placebo for Broccoli Sprout Extract
  Arms: BSE placebo & garlic oil placebo; garlic oil plus BSE placebo
Dietary Supplement: Garlic oil — 1 pill = 30 mg garlic oil/day
  Other Names: Schiff Super Garlic
  Arms: BSE & Garlic Oil; garlic oil plus BSE placebo
Drug: BSE — 2 pills = 200 micromoles of Sulforaphane/day
  Other Names: Broccoli Sprout Extract
  Arms: BSE & Garlic Oil; BSE plus garlic oil placebo
Dietary Supplement: Garlic Oil Placebo — 1 pill = 0 mg garlic oil/day
  Other Names: Placebo for Schiff Super Garlic
  Arms: BSE placebo & garlic oil placebo; BSE plus garlic oil placebo

SUMMARY:
This pilot, three-week study will help scientists understand more about how the foods people eat can modify histone deacetylases, enzymes the body produces naturally. Broccoli sprout extract (BSE) and garlic oil are thought to modify these enzymes. The purpose of this study is to see if taking broccoli sprout extract alone, garlic oil alone, or broccoli sprout extract and garlic oil together, can decrease the action of histone deacetylase (HDAC) and turn on genes in white blood cells. There will be 80 people in this study.

DETAILED DESCRIPTION:
Study participants attend a pre-study meeting either individually or with several other potential volunteers according to their preference. The study is described in detail and participants are given the opportunity to ask questions. If participants agree to participate, they will sign the consent form. Height and weight will be measured privately.

Food diary forms will be distributed and taught how to use. A 4ml (1 tsp) blood sample will be drawn for a pre-study blood chemistry, CBC and thyroid tests. Samples for all clinical labs done during the study will be sent to Good Samaritan Hospital, a CLIA-certified laboratory, on a fee-for-service basis.

The study MD will evaluate the lab results. If the tests are abnormal as determined by the study MD, the participant will be excluded from the study and advised to see their doctor for evaluation.

Subjects will observe dietary restrictions starting one week before Day 1 of the study and continuing through Day 14 (total of 3 weeks). Dietary restrictions are listed on the last page of the diet recall forms.

Women with negative urine pregnancy test on the morning of Day 1 will be enrolled in the study. About 20 ml fasting blood will be drawn on the morning of Day 1. Breakfast will be provided and 3 capsules given to swallow. (One capsule will be garlic oil or garlic oil placebo, the other two will be BSE or BSE placebo.) No eating or drinking (except water) until the next blood draws at 1,3 6 hours after breakfast.

Participants will come to the study site for the next seven days to consume the standard breakfast and study capsules, or we may send the breakfast and study capsules home with participants for the weekend. Blood will be sampled immediately before breakfast on day 7 and again at 1, 3, 6, 24 and 48 hours later. We will provide a standardized lunch to all participants on Days 1 and 7. Additional blood draws will occur at the end of week 2 (i.e. on day 14 of the study). The study will end after 2 weeks.

Participants will fill out a dietary recall form three random times during the study on two week days and one weekend day.

Urine will be collected on the following schedule: Day 1, 0-3 hours, 3-6 hours, 6-12 hours,12-24 hours, 24-48 hours; Day 7, 0-3 hours, 3-6 hours, 6-12 hours, 12-24 hours, 24-48 hours. Total urine from each interval will be collected and pooled in separate containers. We will provide the proper containers for urine collection. Urine may be stored at room temperature.

ELIGIBILITY:
Inclusion criteria:

* age: 20 and older
* body mass index 19-30 kg/sq m
* willingness to maintain normal exercise and activity patterns
* willingness to avoid cruciferous vegetables and garlic and related foods (onion etc.) 1 week before and 2 weeks during the trial for a total of 3 weeks

Exclusion criteria:

* tobacco use within the past three months
* engaging in aerobic activity more than 6 hours per week
* being vegetarian or having other restrictive dietary requirements
* consuming >3 alcoholic beverages/day or >10 per week
* having history of diabetes or uremia or other known metabolic disease
* participating in another dietary study within the past three months
* for women, being pregnant or breastfeeding
* gastrointestinal diseases that could increase gut permeability, including Crohn's disease, ulcerative colitis, gastritis
* taking dietary supplements other than those given in the study
* abnormal liver function, CBC, or thyroid values
* individuals taking any drug or medication, prescription or over the counter, including Isoniazid, Saquinavir, Warfarin, Cyclosporine, Acetaminophen, Oxazepam, medications used for HIV/ AIDS, blood clotting, birth control pills, fish oil and medications metabolized by CYPs (CYP1A2, CYP2E1 and CYP3A4) during the dosing period of 1 week and 48 h prior to and after dosing. Exceptions may be made by the study MD and the PI if in their opinion a medication will not interfere with the scientific validity of the study. The study MD will evaluate a medication on a case-by-case basis to determine that efficacy and safety are not adversely affected.
* Individuals who are known to have problems with blood clotting or increased bleeding, including hemophiliacs or anyone recently undergoing or recovering from a surgical procedure.
* soy or garlic allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Dashwood, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

REFERENCES:
- [Result] Rajendran P, Dashwood WM, Li L, Kang Y, Kim E, Johnson G, Fischer KA, Lohr CV, Williams DE, Ho E, Yamamoto M, Lieberman DA, Dashwood RH. Nrf2 status affects tumor growth, HDAC3 gene promoter associations, and the response to sulforaphane in the colon. Clin Epigenetics. 2015 Sep 18;7(1):102. doi: 10.1186/s13148-015-0132-y. eCollection 2015. PMID 26388957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 Subjects consented for the study at the Linus Pauling Institute clinic, Corvallis, Oregon during the period February, 2013 to November, 2013. However, only 23 who qualified the criteria in the pre-screen blood tests were selected for the study.
Groups:
- BSE Placebo & Garlic Oil Placebo: Two BSE placebo capsules and one garlic oil placebo capsule per day for seven days
  BSE placebo & garlic oil placebo: see arm description
  BSE & Garlic Oil: see arm description
- Garlic Oil Plus BSE Placebo: one garlic oil capsule plus 2 BSE placebo capsules per day for seven days
  BSE placebo & garlic oil placebo: see arm description
  BSE plus garlic oil placebo: see arm description
- BSE Plus Garlic Oil Placebo: two BSE capsules plus one garlic oil placebo capsule per day for seven days
  garlic oil plus BSE placebo: see arm description
  BSE & Garlic Oil: see arm description
- BSE & Garlic Oil: two BSE and one garlic oil capsule per day for seven days
  garlic oil plus BSE placebo: see arm description
  BSE plus garlic oil placebo: see arm description
Period: Overall Study
Arm/Group | BSE Placebo & Garlic Oil Placebo | Garlic Oil Plus BSE Placebo | BSE Plus Garlic Oil Placebo | BSE & Garlic Oil
Started | 5 | 7 | 5 | 6
Completed | 5 | 7 | 5 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BSE Placebo & Garlic Oil Placebo | Garlic Oil Plus BSE Placebo | BSE Plus Garlic Oil Placebo | BSE & Garlic Oil | Total
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (14.1) | 29.9 (10.1) | 30.8 (17.2) | 33.7 (18.1) | 30 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 1 | 12
  Male | 1 | 4 | 1 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 5 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Sulforaphane and Its Metabolites in Blood
Description: The levels of "Sulforaphane and its metabolites (combined)" in blood was measured using Liquid Chromatrography-Mass Spectrometry (LC-MS) methods. Cmax (mean +/- SD) values are shown in the "Outcome Measure Data Table".
Time Frame: Before breakfast (0 hours) and 1, 3 and 6 hours after breakfast & pills on Days 1 & 7, and before breakfast on Days 8, 9 and 14.
Measure: Mean (Standard Deviation); unit: micromoles/L
Arm/Group | BSE Placebo & Garlic Oil Placebo | Garlic Oil Plus BSE Placebo | BSE Plus Garlic Oil Placebo | BSE & Garlic Oil
Number analyzed (Participants) | 5 | 7 | 5 | 6
micromoles/L | NA (NA) — below limit of detection | NA (NA) — below limit of detection | 0.92 (0.15) | 1.26 (0.17)

2. Primary Outcome: Tmax of Sulforaphane and Its Metabolites in Blood
Description: The levels of "Sulforaphane and its metabolites (combined)" in blood was measured using Liquid Chromatrography-Mass Spectrometry (LC-MS) methods. The time to achieve highest plasma concentration (Tmax) is shown in the "Outcome Measure Data Table".
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BSE Placebo & Garlic Oil Placebo | Garlic Oil Plus BSE Placebo | BSE Plus Garlic Oil Placebo | BSE & Garlic Oil
Number analyzed (Participants) | 5 | 7 | 5 | 6
hours | NA (NA) — below limit of detection | NA (NA) — below limit of detection | 3 (0) | 3 (0)

3. Secondary Outcome: Histone Acetylation
Description: Histone acetylation was measured by immunoblotting the levels of acetylated histone H4K12 in the circulating peripheral blood mononuclear cells (PBMCs) of subjects who consumed either placebo, garlic oil, BSE, or BSE+garlic oil. The fold increase in acetylated histone H4K12 in the different groups is shown in the "Outcome Measure Data Table".
Time Frame: 6 h
Population: The data were obtained by analyzing 'representative' patient samples (n=3 per group) using immunoblotting.
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | BSE Placebo & Garlic Oil Placebo | Garlic Oil Plus BSE Placebo | BSE Plus Garlic Oil Placebo | BSE & Garlic Oil
Number analyzed (Participants) | 3 | 3 | 3 | 3
Fold change | 0.83 (0.15) | 1.03 (0.15) | 1.05 (0.21) | 1.20 (0.26)

ADVERSE EVENTS:
Arm/Group | BSE Placebo & Garlic Oil Placebo | Garlic Oil Plus BSE Placebo | BSE Plus Garlic Oil Placebo | BSE & Garlic Oil
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 1/7 | 3/5 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BSE Placebo & Garlic Oil Placebo (N=5) | Garlic Oil Plus BSE Placebo (N=7) | BSE Plus Garlic Oil Placebo (N=5) | BSE & Garlic Oil (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination (23/80) due to small numbers of subjects recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes